CLINICAL TRIAL: NCT03412994
Title: A Randomized, Parallel-controlled, Exploratory Clinical Trial of Second-line Chemotherapy With Second-line Chemotherapy Versus Second-line Chemotherapy With Apatinib in the Treatment of Metastatic Colorectal Cancer
Brief Title: Clinical Study of Apatinib Combined With Second - Line Chemotherapy for Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liqiang Zhong (Other)
Responsible Party: Sponsor-Investigator, Liqiang Zhong, deputy director of the physicians, The Second People's Hospital of Yibin
Organization: The Second People's Hospital of Yibin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR1800014478
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib group (Experimental): Apatinib combined with second-line chemotherapy (5-Fu combined with irinotecan or oxaliplatin standard regimen ) Apatinib tablets: 500 mg po qd . Continuous medication, the cycle is consistent with the chemotherapy cycle.
  Oxaliplatin: Day 1, 130mg/m2, IV infusion. Capecitabine: Day 1-14, 1000mg/m2 Twice Daily, po. A total of 6 cycles, 3 weeks apart of chemotherapy.（Take CAPEOX for example）
  Interventions: Drug: Apatinib; Drug: standard second-line chemotherapy
- Control group (Placebo Comparator): Oxaliplatin: Day 1, 130mg/m2, IV infusion. Capecitabine: Day 1-14, 1000mg/m2 Twice Daily, po. A total of 6 cycles, 3 weeks apart of chemotherapy.（Take CAPEOX for example）
  Interventions: Drug: standard second-line chemotherapy

INTERVENTIONS:
Drug: Apatinib — Apatinib in combination with standard second-line chemotherapy for advanced colorectal cancer
  Other Names: YN968D1
  Arms: Apatinib group
Drug: standard second-line chemotherapy — The second line standard chemotherapy regimen recommended by the NCCN
  Other Names: FOLFOX、FOLFIRI、CapeOX

SUMMARY:
(1) Evaluate the efficacy of apatinib in combination with standard second-line chemotherapy for advanced colorectal cancer. Whether it can prolong Progression Free Survival (PFS), overall survival (OS) in patients with advanced colorectal cancer and reduce symptoms and improve quality of life compared with standard second-line chemotherapy; (2) Observe the safety of apatinib for the treatment of advanced colorectal cancer.

DETAILED DESCRIPTION:
Standard second line chemotherapy includes chemotherapy based on irinotecan or chemotherapy based on oxaliplatin.

Apatinib is a small-molecule tyrosine kinase inhibitor (TKI) that highly selectively binds to and strongly inhibits vascular endothelial growth factor receptor 2 (VEGFR-2), with a decrease in VEGF-mediated endothelial cell migration, proliferation, and tumor microvascular density. A phase II trail of Apatinib has been demonstrated that Apatinib is safe to treat the metastatic colorectal cancer and the disease control rate can reach 50%.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 70 years old;
2. Histologically or cytologically proven patients with metastatic colorectal cancer have undergone a first-line standard regimen recommended by the NCCN guidelines for progression;
3. According to the RECIST 1.1 criteria, the patient has at least one target lesion that can measure the diameter;
4. ECOG PS ≤ 2;
5. Expected survival time of more than 12 weeks.
6. The level of organ function must meet the following requirements:

   Bone marrow: neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelet ≥ 75 × 10^9/L, hemoglobin ≥ 90g/L.

   Liver: serum bilirubin ≤ 2 times the upper limit of normal, aminotransferase AST and ALT ≤ 2.5 times the normal upper limit.

   Kidney: Serum creatinine ≤1.5 times upper limit of normal.
7. Patient compliance is good;
8. Understand and voluntarily sign a written informed consent.

Exclusion Criteria:

1. Other previous or concurrent malignancy, except cured skin basal cell carcinoma and cervical carcinoma in situ;
2. Already known to be allergic to apatinib or any excipient;
3. Use unapproved drugs or other test medications within 4 weeks prior to enrollment;
4. There are many factors that affect oral medications (such as inability to swallow, chronic diarrhea and intestinal obstruction);
5. Patients with a history of CNS metastases or CNS metastases;
6. A history of bleeding, with any serious grading within 4 weeks prior to screening reaching a bleeding event of 3 degrees Celsius or greater in CTCAE4.0;
7. Serious infection;
8. Serious cardiovascular disease: uncontrolled hypertension, unstable angina, grade 3-4 heart failure (NYHA standard), congestive heart failure;
9. urinary routine urinary protein ≥ ++ and confirmed 24-hour urinary protein quantitation> 1.0 g;
10. Within 30 days after major surgery;
11. Thrombotic disease. Anemia or venous thrombosis occurred in the previous year, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, pulmonary embolism, etc.;
12. Those with history of psychotropic substance abuse who can not be abstinent or have mental disorders;
13. Have clinical symptoms, need clinical intervention pleural effusion or ascites;
14. At the investigator's discretion, there is a serious concomitant condition that compromises the patient's safety or affects the patient in completing the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-28 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 2 year
  the time from randomize to progression or death; RECIST guidelines were used to define all responses after patients had received every 4 weeks of therapy

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 3 years
  Defined as the time from randomize to death
Objective Response Rate (ORR) | Approximately 2 years
  ORR=complete response (CR) + partial response (PR)
Disease control rate(DCR) | Approximately 2 years
  Defined as the rate of complete response , partial response and stable disease according to RECIST guidelines
Quality of life(QoL) | Approximately 2 year
  As measured by the European Organization for Research and Treatment of Cancer questionnaire (EORTC QLQ C30)

CONTACTS AND LOCATIONS:
Overall Officials: Liqiang Zhong, Study Chair — Yibin Second People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided